CLINICAL TRIAL: NCT00446355
Title: Clinical Outcomes of Patients With Clostridium Difficile Associated Disease Attributable to Diverse tcdC Genotypes
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Scott Curry, MD, University of Pittsburgh Medical Center
Other Study IDs: PRO07010069
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Clostridium Infections
Keywords: C diff; antibiotics
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to establish the clinical disease outcomes and features of CDAD associated with variant tcdC genotypes. Two hypotheses are to be tested in this study:

1. Severe CDAD and tcdC truncation:

   Severe CDAD (defined by death and/or colectomy or secondary endpoints) is associated with severe truncations (> 6 amino acid residues) in TcdC, a negative regulator of toxin A/B production.
2. Disease in low risk populations (patients never exposed to health care facilities and/or patients who never received antibiotics) of any severity is attributable to strains of C. difficile with severe tcdC truncation.

DETAILED DESCRIPTION:
The following information will be collected: age, sex, occupation, hospital location at the time of positive culture (ER, medical ward, ICU etc), prior hospitalization, receipt of outpatient dialysis, home care or other regular medical care (eg, outpatient chemotherapy), date of specimen collection, presence of invasive devices, receipt of antibiotics, including their type and whether they were adequate for the resistance profile of the organism, prior positive microbiologic cultures, time and location of positive cultures, underlying diseases and severity of illness, presence of urinary or intravascular devices, recent immunomodulative therapies or radiation therapy, physical exam findings, laboratory and radiographical data, antimicrobial usage within 6 months of onset of the infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome,gender, height, weight, ethnicity, past medical history and outcomes. We will collect information retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have confirmed CDAD, confirmed by testing at UPMC's clinical microbiology lab in March 1, 2001- December 31, 2005 for C. difficile by stool toxin test with subsequent positive culture for the organism from inpatients/outpatients at UPMC Presbyterian-Montefiore, from WPIC inpatient units, from ER visits at the Presbyterian University Hospital emergency department, and from clinics closely affiliated with UPMC Presbyterian (medical and surgical clinics in Falk Clinic, the 9 South Montefiore internal medicine clinic, the geriatrics clinic in Montefiore, and the digestive disorders center (GI clinic on 3rd floor of PUH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CDAD confirmed
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Curry, MD, Principal Investigator — University of Pittsburgh; Lee Harrison, MD, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States